CLINICAL TRIAL: NCT07068581
Title: Effect of Maternal Voice on Physiological Indicators and Feeding Performance During Full Oral Feeding Transition in Preterm Infants: A Randomized Controlled Trial
Brief Title: Effect of Maternal Voice on Physiological Indicators and Feeding Performance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Semra Küçük, Research Assistant, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ATADEK-2025/09
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Preterm; Oral Feeding Performance
Keywords: Preterm infants; Oral feeding performance; Maternal voice; NICU care
MeSH Terms: conditions — Premature Birth | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maternal voice group (Experimental): The maternal voice will be played twice daily, starting 20 minutes before the morning and evening oral feedings and continuing throughout the feeding session.
  Interventions: Procedure: Maternal voice
- Standard feeding group (Other): This group will not be exposed to maternal voice before or during feeding; standard feeding care will be provided.
  Interventions: Other: Control Group (standard feeding )

INTERVENTIONS:
Procedure: Maternal voice — Mothers of the infants in the intervention group will be asked to read aloud the lyrics of a designated in a calm tone of voice in a quiet environment, and their voices will be recorded. The recorded maternal voice will then be played to the infants in the NICU using the same Bluetooth-enabled device with built-in speakers. The audio device will be placed inside the incubator or open warmer, approximately 20-30 cm from the infant.
  Each infant will be assigned an individual audio device, which will be used exclusively for that infant. Maternal voice playback will begin 20 minutes before morning and evening oral feedings and will continue throughout the feeding session, twice daily, for a maximum of 5 days. If the infant is discharged earlier, the intervention will be discontinued.. During the playback of the maternal voice, monitor sounds in the NICU will be minimized, and the staff will be instructed to speak quietly to maintain a calm environment.
  Arms: Maternal voice group
Other: Control Group (standard feeding ) — The control group will not be exposed to maternal voice, and standard feeding procedures will be applied.
  Arms: Standard feeding group

SUMMARY:
This study aimed to determine the effect of maternal voice on physiological indicators and oral feeding performance in preterm infants.

Hypothesis 1 (H1): Preterm infants who listen to their mother's voice throughout the full oral feeding process have higher oxygen saturation levels than those who do not.

Hypothesis 2 (H2): Preterm infants who listen to their mother's voice throughout the full oral feeding process have lower heart rates than those who do not.

Hypothesis 3 (H3): Preterm infants exposed to maternal voice throughout the full oral feeding process have lower respiratory rates than those who are not exposed.

Hypothesis 4 (H4): Preterm infants exposed to maternal voice throughout the full oral feeding process have better feeding maturation than those who are not exposed.

Hypothesis 5 (H5): The percentage of nutrient intake in preterm infants exposed to maternal voice throughout the entire oral feeding process is higher than in those not exposed.

Hypothesis 6 (H6): The feeding time of preterm infants exposed to the mother's voice throughout the entire oral feeding process is shorter than that of those not exposed.

Hypothesis 7 (H7): The amount of food consumed per minute by preterm infants exposed to the mother's voice throughout the entire oral feeding process is greater than that of those not exposed.

DETAILED DESCRIPTION:
Oral feeding is one of the critical milestones in the growth and development of preterm infants. A delay in achieving successful oral feeding skills may lead to prolonged hospitalization, negatively impact mother-infant bonding, result in long-term feeding difficulties, impair growth and development, and cause adverse neurodevelopmental outcomes. The literature reports that various methods have been used to enhance oral feeding performance, one of which is maternal voice. It has been reported that the maternal voice has a positive effect on the oral feeding performance of preterm infants. Continuing maternal vocal stimulation during the postnatal period (such as singing lullabies, reading books, or engaging in everyday speech) contributes to strengthening synaptic connections in the auditory cortex, increasing the brain's sensory processing capacity, reducing the infant's stress levels, and maintaining physiological stability. The maternal voice positively influences oral feeding performance by helping infants maintain an alert state and facilitating the coordination of sucking, swallowing, and breathing. In this regard, the maternal voice can be used as an evidence-based nursing intervention to enrich the care of preterm infants. However, the number of high-level evidence studies investigating the relationship between maternal voice and oral feeding performance is limited in the literature, and some existing studies report inconclusive results. Therefore, addressing this issue will help fill a gap in the literature.

In this study, preterm infants in the experimental group will listen to a lullaby recorded in their own mother's voice before and during oral feeding, twice daily (morning and evening) for five consecutive days. A Bluetooth-enabled, speaker-equipped voice recorder will be used for each infant individually. No auditory intervention will be applied to the infants in the control group. In both groups, physiological indicators and oral feeding performance will be measured on specific days.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born at gestational age ≥28 weeks and ≤34 weeks
* Infants who are ≥30 postmenstrual weeks old at the time of enrollment
* Infants weighing ≥1000 grams at the time of enrollment
* Mothers aged 18 years or older
* Preterm infants who have passed the hearing screening test
* Infants whose mothers can provide an average of at least 30 ml of expressed breast milk daily during the study period.
* Mothers who are Turkish speakers.
* Infants for whom the decision to transition from enteral feeding to full oral feeding has been made for the first time jointly by the physician and nurse

Exclusion Criteria:

* Preterm infants with congenital anomalies.
* Infants with a family history of congenital hearing loss.
* Infants diagnosed with intraventricular hemorrhage (grade 3-4) or -periventricular leukomalacia.
* Infants who have had necrotizing enterocolitis requiring treatment.
* Infants whose mothers have a history of substance abuse or alcoholism

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-08-10 (Actual); Primary Completion 2026-07-23 (Estimated); Study Completion 2026-07-23 (Estimated)

PRIMARY OUTCOMES:
Change in Oral Feeding Performance | The first day the infant transitions to full oral feeding and the 5th day will be evaluated. The change between these time points will be assessed.
  Oral feeding performance will be measured using the 'Oral Feeding Maturation Monitoring Device.' One of the device's sensors is positioned under the infant's chin, and the other is placed on the chest. The device evaluates the infant's sucking-swallowing-breathing coordination during a 2-minute feeding session.
Change in oxygen saturation | Oxygen saturation will be measured once daily for five days. Data will be collected immediately before, during, immediately after feeding. The change in these time intervals will be assessed.
  Preterm infant will be monitored and oxygen saturation will be monitored.
Change in heart rate | Heart rate will be measured once daily for five days. Data will be collected immediately before, during, immediately after feeding. The change in these time intervals will be assessed.
  Preterm infant will be monitored and heart rate will be monitored.
Change in respiratory rate | Respiratory rate will be measured once daily for five days. Data will be collected immediately before, during, immediately after feeding. The change in these time intervals will be assessed.
  Preterm infant will be monitored and respiratory rate will be monitored.
Change in Oral Feeding Skills | The first day the infant transitions to full oral feeding and the 5th day will be evaluated. The change between these time points will be assessed.
  Change in oral feeding skills will be assessed using the Early Feeding Skills Assessment Scale.
  The scale was originally developed in 2005, and its Turkish validity and reliability were established in 2021.
  It consists of 5 subdimensions and a total of 19 items. Each item is rated on a scale from 1 to 3. The total score ranges from 19 to 57, with higher scores indicating more advanced feeding skills.

CONTACTS AND LOCATIONS:
Overall Officials: Semra Küçük, Research Assistant,Phd Student, Principal Investigator — Acibadem University
Locations (1):
- Acibadem University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamm EL, Chorna OD, Stark AR, Maitre NL. Feeding outcomes and parent perceptions after the pacifier-activated music player with mother's voice trial. Acta Paediatr. 2015 Aug;104(8):e372-4. doi: 10.1111/apa.13030. Epub 2015 May 16. No abstract available. PMID 25892736
- [Background] Chorna OD, Slaughter JC, Wang L, Stark AR, Maitre NL. A pacifier-activated music player with mother's voice improves oral feeding in preterm infants. Pediatrics. 2014 Mar;133(3):462-8. doi: 10.1542/peds.2013-2547. Epub 2014 Feb 17. PMID 24534413
- [Background] Chirico G, Cabano R, Villa G, Bigogno A, Ardesi M, Dioni E. Randomised study showed that recorded maternal voices reduced pain in preterm infants undergoing heel lance procedures in a neonatal intensive care unit. Acta Paediatr. 2017 Oct;106(10):1564-1568. doi: 10.1111/apa.13944. Epub 2017 Jul 5. PMID 28580602
- [Background] Chhikara A, Hagadorn JI, Lainwala S. Effect of maternal voice on proportion of oral feeding in preterm infants. J Perinatol. 2023 Jan;43(1):68-73. doi: 10.1038/s41372-022-01493-4. Epub 2022 Aug 18. PMID 35982244
- [Background] Alabbasi Y, Parker L, Weaver M, Krueger C. Maternal Voice Exposure and Its Effect on Premature Infants' Feeding Milestones: A Systematic Review. Adv Neonatal Care. 2023 Apr 1;23(2):E40-E49. doi: 10.1097/ANC.0000000000001029. Epub 2022 Oct 3. PMID 36191331